CLINICAL TRIAL: NCT05517473
Title: Efficacy and Safety Evaluation of MONOBLUE DUAL View and MONOBLUE ILM View Vital Stains During Vitrectomy Surgery
Brief Title: Efficacy and Safety Evaluation of MONOBLUE DUAL View and MONOBLUE ILM View Vital Stains
Acronym: NewBlueDyes
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S65841
Record Dates: First submitted 2022-08-18; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Macular Holes; Macular Pucker; Vitreomacular Traction
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators aim to collect data regarding the efficiency and safety of two dyes used intraoperatively in vitrectomy to stain intraocular tissues. These products have the necessary approvals to use during such operation,These are NOT experimental products.

DETAILED DESCRIPTION:
To determine efficacy and safety of MONOBLUE DUAL View and MONOBLUE ILM View (study products) vital stains during vitrectomy surgery.

Both study products are CE-marked and legally marketed in Europe. The data collection will serve as Post-Marketing Clinical Follow-up according MDR provisions. Retrospective data will also be collected for the two reference products: ILM Blue® (DORC) and Membrane Blue Dual® (DORC) to serve as control. For this purpose, patient data will be used that were collected in studies S61408 (Comparative study 23G vs 27G vitrectomy), S63610 (Comparative study 27G vitrectomy vs larger gauge surgery) and S64913 (EVA Nexus Field Observation Study).

The expected effect of the study products is to provide the retinal surgeon with adequate aid in visualizing the membranes involved in the retinal pathology to treat, thanks to their staining capabilities.

The performance of the study products is related to the visualization of retinal tissues (ILM and/or ERM) during the vitrectomy procedure, when these tissues cannot be distinguished accurately enough without staining. Their use allows for better identification of these tissues and facilitates their removal by the surgeon. The clinical benefit of using ophthalmic dyes is to increase the patient's ability to recover anatomically and functionally by allowing more precise surgery with an effective visualization tool.

Along with collecting post-marketing clinical follow-up data on the subject products, the outcomes of the present study results may be used at the UZLeuven Hospital to decide to use Monoblue ILM View and/or Monoblue Dual View as standard-of-care, replacing Membrane Blue Dual and ILM Blue.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who underwent for vitrectomy surgery where ILM and/or ERM removal is required:

* Macular holes (ILM staining)
* Macular pucker (ILM and ERM staining)
* Vitreomacular traction (ILM staining)

Exclusion Criteria:

* Children aged <18 years
* Vitrectomy for other indication than mentioned in 3.1
* Patients that have concomitant eye disease that may influence the outcome of the surgery, e.g. terminal glaucoma
* Patients that did to comply to the postoperative examination visit 6-10 weeks after the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent for vitrectomy surgery where ILM and/or ERM removal is required:
  * Macular holes (ILM staining)
  * Macular pucker (ILM and ERM staining)
  * Vitreomacular traction (ILM staining)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
visualization of membranes | intraoperative (surgery day)
  visualization of membranes stained based on binary subjective evaluation.

SECONDARY OUTCOMES:
surgical help | intraoperative (surgery day)
  subjective assessment of surgical help provided by the product
adverse events | 1 day after surgery
  Rate and severity of potential study-related products adverse events
visual acuity | 6 weeks after surgery
  Visual outcome at the last postoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, Phd, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT05517473/Prot_SAP_000.pdf